CLINICAL TRIAL: NCT01371188
Title: Effects of Exposure to Outdoor Air Pollution From Biomass Burning on Lung Function, Heart Rate Variability and Systemic Inflammatory Blood Markers in Sugarcane Workers
Brief Title: Effects of Exposure to Biomass-burning Air Pollution on Lung Function, Heart Rate Variability and Inflammatory Markers in Sugarcane Workers
Status: Completed | Type: Observational
Sponsor: InCor Heart Institute (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Dr Ubiratan de Paula Santos and Dr. Gustavo Faibischew Prado, InCor
Other Study IDs: Mendonca; 402195/2008 (Other: CNPQ)
Record Dates: First submitted 2011-06-09; First posted 2011-06-10 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-06

CONDITIONS: Lung Function; Heart Rate Variability; Oxidative Stress; Systemic Inflammatory Response

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Controls: Healthy male volunteers, non-smokers, 20-40yo, living in the city of Mendonça, São Paulo-Brazil.
- Sugarcane Workers: Healthy male volunteers, non-smokers, 20-40yo, sugarcane workers, living in the city of Mendonça, São Paulo-Brazil.

SUMMARY:
Introduction: Non-mechanized sugar cane harvesting preceded by burning, an important and prevalent professional activity of agribusiness segment of the Brazilian economy, exposes workers and people of neighboring towns to high concentrations of pollutants and, therefore, potentially several risks to health hazards.

Objectives: Assessing cardiopulmonary impacts and inflammatory markers in sugarcane workers and volunteers from a nearby town in non-harvest and harvest periods.

ELIGIBILITY:
Inclusion Criteria:

* The criteria for inclusion in the study were: age between 20 and 40 years, male gender and being non-smokers (or former-smokers for at least a year and a smoking history of less than 20 pack-years).

Exclusion Criteria:

* Exclusion criteria were history of cardiovascular or respiratory disease, the use of bronchodilator, non-steroidal anti-inflammatory drugs, anticoagulants or antiplatelet drugs and statins.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Population from the city of Mendonça, São Paulo-Brazil, divided into the following groups: sugarcane workers (those who work in sugarcane plantations) and controls (healthy volunteers from the same city)
Sampling Method: Non-Probability Sample
Enrollment: 222 (Actual)
Dates: Start 2008-12; Primary Completion 2010-10 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Lung function | six months
  Measurements of lung function in pre harvest and during harvest period
Heart rate variability | six months
  To evaluate parameters of heart rate variability in pre harvest and during harvest periods
Oxidative stress | six months
  Measurement of blood levels of antioxidant enzymes and malonaldehyde

SECONDARY OUTCOMES:
Environmental evaluation | one year
  Measurement of athmospheric concentration of particulate matter.

CONTACTS AND LOCATIONS:
Locations (1):
- City of Mendonça (urban area and sugarcane plantations), Mendonça, São Paulo, Brazil

REFERENCES:
- [Derived] Paula Santos U, Zanetta DM, Terra-Filho M, Burdmann EA. Burnt sugarcane harvesting is associated with acute renal dysfunction. Kidney Int. 2015 Apr;87(4):792-9. doi: 10.1038/ki.2014.306. Epub 2014 Sep 17. PMID 25229334